CLINICAL TRIAL: NCT03625193
Title: Appropriate Methods and Psychometric Properties of Sit-to-stand Test in Ambulatory Patients With Spinal Cord Injury
Brief Title: Psychometric Properties of Sit-to-stand Test in Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sugalya Amatachaya, Assoc. Prof. Dr., Khon Kaen University
Other Study IDs: PHD02232558
Record Dates: First submitted 2018-01-10; First posted 2018-08-10 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2018-08

CONDITIONS: Spinal Cord Injuries
Keywords: Sit-to-stand test; Psychometric properties
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ambulatory patients with SCI: * Age at least 18 years
  * Body mass index (BMI) between 18.5 - 29.9 kg/m2
  * Having an incomplete SCI from traumatic or non-traumatic causes
  * Ability of independent standing up from a chair with or without hand support
  * Ability of independent walking with or without walking device over at least 10 meters continuously.
  * Ability to follow commands used in the studies

SUMMARY:
1. Do different arm placements (including arms on armrests/devices, arms on knees, arms free, and arm crossed over chest) influence outcomes of sit-to-stand test (STST) in ambulatory individuals with spinal cord injury (SCI)?
2. What are the factors associated with ability to perform STST in ambulatory individuals with SCI?
3. Are the single-time sit-to-stand test (STSST) and five-time sit-to-stand test (FTSST) reliable, valid and responsive to determine functional alteration in ambulatory individuals with SCI?

DETAILED DESCRIPTION:
* To cross-sectionally compare characteristics (duration and amount of lower limb loading) of STS movements among 4 arm placement conditions (arms on armrests/devices, arms on knees, arms free, and arm crossed over chest) in ambulatory patients with SCI.
* To investigate reliability (inter-rater, intra-rater, and test-retest), standard error of measurement and minimal detectable changes of the STSST and FTSST in ambulatory patients with SCI.
* To investigate concurrent validity and factors associated with ability of the STSST and FTSST in ambulatory patients with SCI.
* To investigate the ability of the STSST and FTSST to predict the risk of falls over 1, 3 and 6 months in ambulatory patients with SCI.
* To investigate internal and external responsiveness of the STSST and FTSST to detect changes on walking ability over 1, 3 and 6 months in ambulatory patients with SCI.
* To estimate the minimal clinically important difference or clinical significance of the FTSST in ambulatory patients with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 - 29.9 kg/m2
* Having an incomplete SCI from traumatic or non-traumatic causes
* Ability of independent standing up from a chair with or without hand support
* Ability of independent walking with or without walking device over at least 10 meters continuously.
* Ability to follow commands used in the studies

Exclusion Criteria:

Any ambulatory individuals with incomplete SCI who present signs and symptoms that might affect ability to perform STST will be excluded from the study such as

* Pain in the muscles or joints with an intensity of pain more than 5 out of 10 on a numeric rating scale (NRS)
* Joint deformities that affect mobility
* Other neurological disorders such as having brain lesions
* Unstable medical conditions
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is conducted in patients with spinal cord injury who able to sit-to-stand independently with or without hand support from the Srinagarind hospital and communities in the Northeast areas of Thailand.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Ability to perform single and five times sit-to-stand test among 4 arm conditions | Change over 6 months
  Ability to execute a single time sit-to-stand and time used for five times sit-to-stand

SECONDARY OUTCOMES:
10-meter walk test | Change over 6 months
  Change in walking speed during 6-month follow-up
Fall events | Over 6 months
  Incidence of fall during 6-month follow-up
Global rating of change score (GRC score) | Change over 6 months
  Level of change in subjects' independence in activities of daily life. The GRC score is divided into 15-point scale from "-7" (a very great deal worse) to "0" (about the same/ not change) to "7" (a very great deal better).

CONTACTS AND LOCATIONS:
Overall Officials: Sugalya Amatachaya, PhD, Principal Investigator — School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Khon Kaen, Thailand.
Locations (1):
- Faculty of Associated Medical Science, 123 Moo 16 Mittapap Rd., Nai-Muang, Muang District, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No